CLINICAL TRIAL: NCT03919643
Title: B Cell Activating Factor Belonging to the TNF (Tumor Necrosis Factor) Family (BAFF) and a Proliferation-inducing Ligand (APRIL) in Patients With Systemic Lupus Erythematosus: Investigating Biomarkers for the Response to the Belimumab Treatment
Brief Title: BAFF and APRIL and RESPONSE TO BELIMUMAB in SLE
Acronym: BAFF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: BAFF
Record Dates: First submitted 2019-02-14; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Systemic Lupus Erythematosus; BAFF Polymorphism
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE patients with nephritis: No intervention. Peripheral blood and urine samples will be obtained
- SLE patients with without nephritis: No intervention. Peripheral blood and urine samples will be obtained
- Healthy controls (blood donors): No intervention. Peripheral blood and urine samples will be obtained

SUMMARY:
This project is intended to identify the routes on which BAFF and APRIL act in order to detect possible future candidates to Belimumab treatment among patients diagnosed of SLE.

DETAILED DESCRIPTION:
DESIGN Establish the influence of certain polymorphisms in the levels of expression of different transcripts and proteins.

Quantify the levels of B cell activating factor belonging to the TNF family (BAFF) and a proliferation-inducing ligand (APRIL) in serum and urine of patients and controls by Enzyme-Linked Immunosorbent Assay (ELISA). BAFF Determine the expression levels of different BAFF and APRIL transcripts in peripheral blood mononuclear cells from patients and controls using a digital PCR (polymerase chain reaction) system.

Compare distribution of gene polymorphisms in BAFF and APRIL in patients and controls. by sequencing the exome of the ligand and receptor genes using next generation sequencing (NGS).

Correlate the transcript and protein levels with clinical manifestations and disease activity.

The results of the quantification of anti- double-stranded deoxyribonucleic acid.(dsDNA) antibody levels tests will be recorded together with those demographics, clinical-epidemiological and response to the treatment.data.

ELIGIBILITY:
Inclusion criteria

* Women18-60 years old
* For patients only treated with conventional drugs (without immunosuppressive or biological treatment )
* For Healthy controls: no autoimmune diseases (blood donors) diagnoses

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SLE (Sistemic Lupus Disease) with and without nephritis and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Improve knowledge of B Cell activating factor belonging to the TNF (Tumor necrosis factor) family (BAAF) system in order to identify those SLE (Systemic Lupus Erythematous) patients that are candidate for treatment with anti-BAFF. | from data of Informed consent form signature to finish of follow-up (1 Year)
  Quantify physiological parameters (levels of BAFF and APRIL) in serum and urine of patients and controls by ELISA.
Establish the influence of certain polymorphisms in the levels of expression of different transcripts and proteins. | from data of Informed consent form signature to finish of follow-up (1 Year)
  Determine the expression levels of different physiological parameters (BAFF and APRIL transcripts) in peripheral blood mononuclear cells from patients and controls.
Correlate the transcript and protein levels with clinical manifestations and disease activity. | from data of Informed consent form signature to finish of follow-up (1 Year)
  Quantify anti-dsDNA levels recording clinical symptoms and SLE-DAI (Systemic Lupus Erythematosus Disease Activity Index)

IPD SHARING:
Plan to Share IPD: Yes
Sharing the data collected and analysed with the scientific community by publication
Supporting Information: Study Protocol, ICF
Time Frame: When study is finished
Access Criteria: Data publication for collaborator, data base registration of results if applicable.

REFERENCES:
- [Derived] Ortiz-Aljaro P, Montes-Cano MA, Garcia-Lozano JR, Aquino V, Carmona R, Perez-Florido J, Garcia-Hernandez FJ, Dopazo J, Gonzalez-Escribano MF. Protein and functional isoform levels and genetic variants of the BAFF and APRIL pathway components in systemic lupus erythematosus. Sci Rep. 2022 Jul 2;12(1):11219. doi: 10.1038/s41598-022-15549-0. PMID 35780200